CLINICAL TRIAL: NCT04563559
Title: Patient PReference, Efficacy, and SaFety of an Intracanalicular DExamenthasone InseRt comparEd to Topical PrednisoloNe in PatienTs UndergoIng SequentiAl PhacoemuLsification With Intraocular Lens Surgery OR Combined Phacoemulsification With IOL and a Minimally Invasive Glaucoma Surgery (MIGS)
Brief Title: PREFERENTIAL Study
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: PI decided not to open study
Sponsor: Duke University (Other)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00104649
Record Dates: First submitted 2020-09-21; First posted 2020-09-24 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Cataract Surgery; Glaucoma Surgery
MeSH Terms: interventions — Calcium Dobesilate; prednisolone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- DEXTENZA vs prednisolone acetate 1%) (Other): Subjects will randomly receive Dextenza or prednisolone acetate 1% in the first eye after surgery. At the time of the second eye surgery, the other eye will receive the drug that the first eye did not receive. Subjects will receive both drugs during the course of the study and therefore there is only 1 ARM for this study.
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert; Drug: Prednisolone Acetate 1% Ophthalmic Suspension [PRED FORTE]

INTERVENTIONS:
Drug: Dextenza 0.4Mg Ophthalmic Insert — The eye will have a sustained release device of Dexamethasone 0.4 mg placed in the inferior nasal lacrimal system.
Drug: Prednisolone Acetate 1% Ophthalmic Suspension [PRED FORTE] — The eye will be randomized to receive topical treatment with prednisolone acetate 1% on a tapering dose schedule

SUMMARY:
To determine patient preference for the dexamethasone insert or topical prednisolone therapy through at Day 45 as measured by - Modified COMTOL survey.

DETAILED DESCRIPTION:
Eyes from 80 patients will be randomized in a 1:1 ratio to the assigned treatment, dexamethasone insert placed at the time of surgery, or topical prednisolone acetate 1% therapy prescribed on a tapering dose schedule post-operatively.

Males and Females 18 years and older with 1)Presence of a visually significant cataract with plans to undergo clear cornea cataract surgery with phacoemulsification and implantation of a posterior chamber intraocular lens (IOL), and potential postoperative Snellen pinhole corrected distance visual acuity (CDVA) of at least 20/200 in both eyes and 2) 10 patients with mild-to-moderate primary open angle glaucoma and a visually significant cataract with plans to undergo clear cornea cataract surgery with phacoemulsification and implantation of a posterior chamber Intraocular Len (IOL) combined with a Minimally Invasive Glaucoma Surgery (MIGS) procedure in both eyes.

Study visits will consist of eye exam with ocular photos from an Optical Coherence Tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Presence of a visually significant cataract with plans to undergo clear cornea cataract surgery with phacoemulsification and implantation of a posterior chamber intraocular lens (IOL), and potential postoperative Snellen pinhole CDVA of at least 20/200 in both eyes
* 10 patients with mild-to-moderate primary open angle glaucoma and a visually significant cataract with plans to undergo clear cornea cataract surgery with phacoemulsification and implantation of a posterior chamber IOL combined with a Minimally Invasive Glaucoma Surgery (MIGS) procedure in both eyes

Exclusion Criteria:

* Active or history of chronic or recurrent inflammatory eye disease in either eye
* Ocular pain in either eye
* Proliferative diabetic retinopathy in either eye
* Significant macular pathology detected on macular optical coherence tomography evaluation at the screening visit in either eye
* Laser or incisional ocular surgery during the study period and 6 months prior in either eye
* Systemic concomitant pain medication management with pharmacologic class of oxycodone
* Systemic NSAID use

  o Pre-procedural wash-out period for topical NSAIDS, ocular steroid, cyclosporine of 7 days
* Clinically significant macular edema (CSME)
* History of cystoid macular edema in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Percent of patients who stated they preferred dexamethasone insert as measured by patient report | 45 days post second surgery
  To determine patient preference for the dexamethasone insert or topical prednisolone therapy through at Day 45 as measured by Modified COMTOL survey.
Percent of patients who stated they preferred topical prednisolone insert as measured by patient report | 45 days post second surgery
  To determine patient preference for the dexamethasone insert or topical prednisolone therapy through at Day 45 as measured by Modified COMTOL survey.

SECONDARY OUTCOMES:
The incidence of AE | Up to 3 months
  The incidence of adverse events
The severity of AE | Up to 3 months
  The severity of adverse events
Resolution of inflammation | Day 14 post surgery
  Resolution of inflammation as defined as either 0 or 0.5 cells or less cells on post-surgical day 14 as measured by SUN scale in an unmasked fashion.
Resolution of pain | Day 7 post surgery
  Resolution of pain as defined by a score of 0 measured by pain scale on post-surgical day 7
Absence of cell flare at day 14 | Day 14 post surgery
  Absence of cell flare at day 14
Mean change in BCVA | Baseline, 3 months
  Mean change in BCVA
Mean change in central retinal thickness as measured by OCT | Baseline, 3 months
  Mean change in central retinal thickness as measured by OCT
Percent of patients who maintained normalized central retinal thickness at 28 days post surgery | 28 days post surgery
  Percent of patients who maintained normalized central retinal thickness at 28 days post surgery
Percent of patients with rebound inflammation | Up to 3 months
  Percent of patients with rebound inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Leon Herndon, MD, Principal Investigator — Duke Eye Center

IPD SHARING:
Plan to Share IPD: No